CLINICAL TRIAL: NCT05431179
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Zilovertamab (an ROR1 Antibody) Plus Ibrutinib Versus Ibrutinib Plus Placebo in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: A Study of Zilovertamab and Ibrutinib in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a strategic reprioritization based on the rapidly changing clinical and commercial landscape for Bruton's tyrosine kinase inhibitors (BTK inhibitors)
Sponsor: Oncternal Therapeutics, Inc (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZILO-301
Record Dates: First submitted 2022-06-09; First posted 2022-06-24 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Lymphoma, Mantle-Cell; Lymphoma; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell
Keywords: Mantle cell lymphoma; Receptor Tyrosine Kinase-like Orphan Receptor 1 (ROR1); Bruton Tyrosine Kinase (BTK) inhibitor; Ibrutinib; Zilovertamab
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — cirmtuzumab; ibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Ibrutinib (Experimental): Open Label Ibrutinib Monotherapy Phase (16 weeks)
  Interventions: Drug: Ibrutinib
- Arm A: IV Infusion of Ziloveramab and Oral Ibrutinib (Experimental): Randomized, Double-Blind Treatment Phase
  Interventions: Drug: Zilovertamab; Drug: Ibrutinib
- Arm B: IV Infusion of Placebo and Oral Ibrutinib (Placebo Comparator): Randomized, Double-Blind Treatment Phase
  Interventions: Drug: Ibrutinib; Drug: Placebo

INTERVENTIONS:
Drug: Zilovertamab — After 16 weeks in the open-label Ibrutinib phase, participants will receive zilovertamab (600mg) administered by IV every 2 weeks for 3 administrations and then every 4 weeks thereafter.
  Other Names: Cirmtuzumab; UC961
  Arms: Arm A: IV Infusion of Ziloveramab and Oral Ibrutinib
Drug: Ibrutinib — All participants will receive oral Ibrutinib (560mg) daily.
  Other Names: Imbruvica
Drug: Placebo — After 16 weeks in the open-label Ibrutinib phase, participants will receive placebo administered by IV every 2 weeks for 3 administrations and then every 4 weeks thereafter.
  Arms: Arm B: IV Infusion of Placebo and Oral Ibrutinib

SUMMARY:
This is a Phase 3 study to investigate the safety and efficacy of the investigational drug, zilovertamab, when given in combination with ibrutinib in patients with relapsed/refractory (R/R) mantle cell lymphoma (MCL).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study that will be conducted in multiple phases in patients with R/R MCL. The study phases will include a Screening Phase, an Open-Label Ibrutinib Monotherapy Treatment Phase, a Randomized Double-Blind Treatment Phase, and a Long-Term Follow-Up Phase. When patients meet all study eligibility requirements in the Screening Phase, they will enter the Open-Label Ibrutinib Monotherapy Treatment Phase and will receive ibrutinib alone daily. After approximately 16 weeks patients who have a partial response (PR) or stable disease (SD) will enter the Randomized Double-Blind Treatment Phase and will be receive an intravenous infusion of zilovertamab or placebo and will continue to receive ibrutinib daily. Patients who discontinue study drug will enter the Long-Term Follow-Up Phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed MCL
* Has received one prior regimen for MCL
* Disease is relapsed or refractory
* At least 1 measurable site of disease that is ≥ 2.0 cm
* PET-CT performed less than 28 days before study entry
* If a subject has toxicities due to prior therapy for the treatment of MCL, must be stable and recovered
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Study-specific laboratory parameters must be met
* Females of childbearing potential and males must use highly effective contraception

Exclusion Criteria:

* Received more than one month of prior therapy with ibrutinib or any other Bruton's tyrosine kinase inhibitor
* Concurrent enrollment in another investigational study
* Transfusion-dependent thrombocytopenia
* Anticancer therapy within 25 days before the start of the study
* History of other malignancy, cancer, or carcinoma for at least three years before the start of the study
* Central nervous system (CNS) involvement with lymphoma
* CNS disorder ≤ 6 months of study entry
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, active arrhythmias, class 3 or 4 congestive heart failure, or other clinically significant cardiac disease ≤ 6 months of study entry
* Active or prior cardiac (atrial or ventricular) lymphoma involvement
* History of atrial fibrillation or left or right bundle branch block
* History of symptomatic deep vein thrombosis or pulmonary embolism ≤ 6 months of study entry
* Chronic liver disease with hepatic impairment, Child-Pugh class B or C
* Bleeding disorder
* Prior stem cell transplant that requires ongoing immunosuppressive therapy or active clinical graft versus host disease
* Primary severe immunodeficiency
* Human immunodeficiency virus infection (HIV) or active hepatitis B or C infection
* Active infection requiring IV antimicrobial (antiviral, antibiotic, anti-fungal) therapy at the time of study entry
* Vaccination with a live, attenuated vaccine ≤ 4 weeks of the start of the study
* Hypersensitivity reaction to any of the agents used in this study
* Requires treatment with a strong cytochrome P450 enzyme (CYP) 3A (CYP3A) inhibitor/inducer.
* Unable or swallow capsules or tablets or has malabsorption syndrome or disease affecting gastrointestinal function
* Major surgery ≤ 4 weeks of study start
* Medical condition likely to interfere with assessment of safety or efficacy of the study drug
* Not eligible in the opinion of the Investigator
* Pregnant or breastfeeding

Other protocol-defined inclusion/exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 2 years
  PFS as assessed by Blinded Independent Central Review (BICR) per Lugano Classification is superior for ibrutinib plus zilovertamab compared to ibrutinib plus placebo among subjects with relapsed or refractory (R/R) mantle cell lymphoma (MCL) that had a PR or SD after 16 weeks of ibrutinib monotherapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 4 years
  Assessed by BICR per Lugano Classification, among the subjects who received the combination of zilovertamab plus ibrutinib compared with the subjects who received ibrutinib plus placebo.
Duration of Response (DOR) | Approximately 4 years
  Assessed by BICR per Lugano Classification, among the subjects who received the combination of zilovertamab plus ibrutinib compared with the subjects who received ibrutinib plus placebo.
Complete Response Rate | Approximately 4 years
  Assessed by BICR per Lugano Classification Classification among the subjects who received the combination of zilovertamab plus ibrutinib compared with the subjects who received ibrutinib plus placebo.
Proportion of subjects experiencing Grade 3 to 4 neutrophil count decrease | Approximately 4 years
  Proportion of subjects experiencing Grade 3 to 4 neutrophil count decrease among the subjects who received the combination of zilovertamab plus ibrutinib compared with the subjects who received ibrutinib plus placebo based on laboratory abnormalities.
Overall Survival (OS) | Approximately 4 years
  OS among the subjects who received the combination of zilovertamab plus ibrutinib compared with the subjects who received ibrutinib plus placebo.
Overall Safety Profile | Approximately 4 years
  Overall safety profile among the subjects who received the combination of zilovertamab plus ibrutinib compared with the subjects who received ibrutinib plus placebo. This would include incidence of treatment-emergent adverse events and laboratory abnormalities.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753